CLINICAL TRIAL: NCT04624503
Title: Prognostic and Clinical Impact of Cardiovascular Involvement in Patients With COVID-19 (Rilevanza Clinica e Prognostica Del Coinvolgimento Cardiovascolare Nei Pazienti Affetti da COVID-19)
Brief Title: Prognostic and Clinical Impact of Cardiovascular Involvement in Patients With COVID-19
Acronym: CARDIO-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Humanitas Hospital, Italy (Other)
Collaborators: Centro Cardiologico Monzino (Other); IRCCS Policlinico S. Donato (Other); Istituti Clinici Scientifici Maugeri SpA (Other); Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Giulio Stefanini, Prof., Humanitas Hospital, Italy
Other Study IDs: CARDIOCOVID
Record Dates: First submitted 2020-10-17; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Myocardial Injury; Cardiovascular Diseases; Heart Failure; Cardiovascular Morbidity
Keywords: Cardiovascular involvement; COVID-19
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 infection has been associated with numerous cardiac manifestations. Indeed, SARS-CoV-2 may impact on cardiovascular system through a direct myocardial infection or a secondary cardiac involvement due to hypoxia or metabolic supply-demand imbalance or prothrombotic inflammatory state. As a consequence of and besides acute myocardial damages, COVID-19 could also determine chronic cardiovascular consequences, with a significant impact on long-term prognosis, quality of life and functional capacity of COVID-19 survivors.

On this basis, we aim to define the clinical and prognostic effects of myocardial involvement in COVID-19 patients.

DETAILED DESCRIPTION:
COVID-19 infection has been associated with numerous cardiac manifestations. Indeed, SARS-CoV-2 may impact on cardiovascular system through a direct myocardial infection or a secondary cardiac involvement due to hypoxia or metabolic supply-demand imbalance or prothrombotic inflammatory state. As a consequence of and besides acute myocardial damages, COVID-19 could also determine chronic cardiovascular consequences, with a significant impact on long-term prognosis, quality of life and functional capacity of COVID-19 survivors.

On this basis, we aim to define the clinical and prognostic effects of myocardial involvement in COVID-19 patients, with a 1-month and 6-month follow-up composed of clinical evaluation, electrocardiogram, trans-thoracic echocardiogram, cardiovascular magnetic resonance, chest computerized tomography scan and cardiopulmonary exercise test.

ELIGIBILITY:
Inclusion Criteria: patients who were hospitalized for COVID-19

Exclusion Criteria: None.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | 1 month
  Mortality due to cardiovascular causes at 1 month after hospitalization
Cardiovascular mortality | 6 months
  Mortality due to cardiovascular causes at 6 months after hospitalization
All-cause mortality | 1 month
  Mortality due to all causes at 1 month after hospitalization
All-cause mortality | 6 months
  Mortality due to all causes at 6 months after hospitalization
Major adverse cardiovascular events (myocardial infarction, cerebrovascular accident, hospitalizations due to heart failure, revascularizations, cardiovascular mortality) | 1 month
  Major adverse cardiovascular events at 1 month after hospitalization
Major adverse cardiovascular events (myocardial infarction, cerebrovascular accident, hospitalizations due to heart failure, revascularizations, cardiovascular mortality) | 6 months
  Major adverse cardiovascular events at 6 months after hospitalization

SECONDARY OUTCOMES:
NYHA class | 6 months
  NYHA functional class: from I (no limitation of physical activity) to IV (severe limitation with symptoms at rest)
Left ventricular systolic function (cardiac magnetic resonance, echocardiography) | 6 months
  Left ventricular systolic function evaluated with multimodality imaging

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Condorelli, Prof, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (5):
- Italy (5):
  - Humanitas Research Hospital, Rozzano, Milan
  - Centro Cardiologico Monzino, Milan
  - IRCCS Auxologico San Luca, Milan
  - IRCCS San Donato, Milan
  - IRCCS Istituti Clinici Scientifici Maugeri, Pavia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stefanini GG, Chiarito M, Ferrante G, Cannata F, Azzolini E, Viggiani G, De Marco A, Briani M, Bocciolone M, Bragato R, Corrada E, Gasparini GL, Marconi M, Monti L, Pagnotta PA, Panico C, Pini D, Regazzoli D, My I, Kallikourdis M, Ciccarelli M, Badalamenti S, Aghemo A, Reimers B, Condorelli G; Humanitas COVID-19 Task Force. Early detection of elevated cardiac biomarkers to optimise risk stratification in patients with COVID-19. Heart. 2020 Oct;106(19):1512-1518. doi: 10.1136/heartjnl-2020-317322. Epub 2020 Aug 14. PMID 32817312